CLINICAL TRIAL: NCT07241715
Title: Conversion Surgery for Gastric Cancer With Peritoneal Metastases (CONVERGENCE)
Acronym: CONVERGENCE
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Karolinska University Hospital (Other); University of Lyon (Other); M.D. Anderson Cancer Center (Other); Seoul National University Hospital (Other); University of Oxford (Other); Peter MacCallum Cancer Centre, Australia (Other); Queen Mary Hospital, Hong Kong (Other); Chinese University of Hong Kong (Other); University Hospital, Lille (Other); Erasmus Medical Center (Other); University Hospital, Montpellier (Other); Universita di Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/00052
Record Dates: First submitted 2024-10-07; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Gastric Cancer Stage IV; Peritoneal Metastasis
Keywords: Gastric cancer; Peritoneal Metastasis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Conversion to Open Surgery; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conversion surgery with systemic therapy (including 1L chemotherapy +/- targeted therapy +/- immunot (Experimental)
  Interventions: Procedure: Conversion Surgery
- systemic therapy (including 1L chemotherapy +/- targeted therapy +/- immunotherapy) +/- peritoneal d (Active Comparator)
  Interventions: Drug: Systemic Therapy/Standard of Care

INTERVENTIONS:
Procedure: Conversion Surgery — Conversion surgery with systemic therapy (including 1L chemotherapy +/- targeted therapy +/- immunotherapy) +/- peritoneal directed chemotherapy
  Arms: Conversion surgery with systemic therapy (including 1L chemotherapy +/- targeted therapy +/- immunot
Drug: Systemic Therapy/Standard of Care — systemic therapy (including 1L chemotherapy +/- targeted therapy +/- immunotherapy) +/- peritoneal directed chemotherapy
  Arms: systemic therapy (including 1L chemotherapy +/- targeted therapy +/- immunotherapy) +/- peritoneal d

SUMMARY:
The goal of this clinical trial is to evaluate the impact of conversion surgery on overall survival (OS) in patients with gastric cancer peritoneal metastases (GCPM) who show a good response to preoperative systemic therapy (including first-line chemotherapy with or without targeted therapy and/or immunotherapy) with or without peritoneal-directed chemotherapy.]. The main question it aims to answer is:

(i) Will Conversion surgery be associated with improved overall survival (OS) in patients with GCPM who respond well to preoperative systemic therapy, compared to patients who do not undergo surgery? (ii) Will Quality of life be comparable or improved in patients who undergo conversion surgery compared to patients receiving palliative chemotherapy as measured by the QLQ-C30 questionnaire?

If there is a comparison group: Researchers will compare Arm 1 (Conversion surgery with systemic therapy (including 1L chemotherapy +/- targeted therapy +/- immunotherapy) +/- peritoneal directed chemotherapy) to Arm 2 (systemic therapy alone (including 1L chemotherapy +/- targeted therapy +/- immunotherapy) +/- peritoneal directed chemotherapy) to see if the conversion surgery will be associated with improved overall survival (OS) in Arm 1.

Participants will be randomized to either Arm 1 or Arm 2.

* For Arm 1, participants will go for conversion surgery then continue systemic therapy.
* For Arm 2, participants will continue systemic therapy.

Radiological assessment will be performed every 6 months or upon progression of disease, whichever comes earlier.

ELIGIBILITY:
Inclusion Criteria:

* GCPM detected on surgical exploration and demonstrated by histology or cytology
* Primary GC not resected
* Age > 21 (or > 18 as allowed by individual institution review boards)

Exclusion Criteria:

* Pregnant and lactating females
* Prior surgical treatment for GC involving resection
* Clinical or radiological progression during 1st line systemic treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2034-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From enrollment to the end of follow-up at 36 months.
  Time from randomization to death from any cause. Patients alive or lost to follow-up at analysis will be censored at the date last known alive.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From enrollment to the end of follow-up at 36 months.
  Time from randomization to radiological or clinical recurrence (Arm 1) or progression (Arm 2), or death from any cause, whichever occurs first. Patients alive and without recurrence/progression will be censored at the date last known disease-free.
Surgical outcomes | From surgery to 90 days post-operation, and up to the end of follow-up at 36 months for late events.
  Incidence of postoperative complications graded according to the Clavien-Dindo classification.
Quality of Life - Global Health Status (EORTC QLQ-C30 | Baseline and scheduled follow-up visits up to 36 months.
  Change in global health status/quality-of-life score using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). Scale 0-100; higher scores indicate better global health/QoL.
Quality of Life - Gastro-Oesophageal Symptoms (EORTC QLQ-OG25) | Baseline and scheduled follow-up visits up to 36 months.
  Change in symptom-specific scores using the EORTC QLQ-OG25 module assessing upper GI symptoms and treatment-related side effects. Scale 0-100; higher scores indicate worse symptoms.
Quality of Life - General Health Status (EQ-5D-5L) | Baseline and scheduled follow-up visits up to 36 months.
  Change in EQ-5D-5L health status index (range -0.594 to 1.0; higher indicates better health) and visual analog scale (VAS 0-100; higher indicates better perceived health).

IPD SHARING:
Plan to Share IPD: Undecided